CLINICAL TRIAL: NCT00275262
Title: Leuprolide Acetate to Enhance Immune Function Post-Autologous Stem Cell Transplantation
Brief Title: A Study to Evaluate the Ability of Lupron Depot to Enhance Immune Function Following Bone Marrow Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Norwood Immunology Limited (Unknown); M.D. Anderson Cancer Center (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Kristof Chwalisz, Therapeutic Area Head, Abbott
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: L-BT04-093
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Results first posted 2010-05-06 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2010-04

CONDITIONS: Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma; Mantle Cell Lymphoma
Keywords: Bone marrow transplantation; Hematopoietic stem cell transplantation; Hodgkin's disease; non-Hodgkin's lymphoma; multiple myeloma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma; Lymphoma, Mantle-Cell | interventions — Leuprolide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LAD 11.25 mg 3 Month Depot (Experimental): Three intramuscular injections LAD 11.25 mg 3 Month treatment administered approximately 3 months apart.
  Interventions: Drug: Leuprolide acetate depot (LAD) 11.25 mg 3 Month
- Placebo Comparator (Placebo Comparator): Three intramuscular injections of matched placebo administered approximately 3 months apart.
  Interventions: Drug: Matched placebo

INTERVENTIONS:
Drug: Leuprolide acetate depot (LAD) 11.25 mg 3 Month — LAD intramuscular injection 11.25 mg, 3 month duration. To stimulate immune response, a subcutaneous key limpet hemocyanin (KLH) vaccination injection (1 mg) was administered at Month 6.
  Other Names: Lupron
  Arms: LAD 11.25 mg 3 Month Depot
Drug: Matched placebo — Matched placebo intramuscular injection, 3 month duration. To stimulate immune response, a subcutaneous key limpet hemocyanin (KLH) vaccination injection (1 mg) was administered at Month 6.
  Arms: Placebo Comparator

SUMMARY:
Phase 2 study, conducted in patients with Hodgkin's disease, non-Hodgkin's lymphoma, multiple myeloma, or mantle cell lymphoma undergoing high-dose chemotherapy and autologous stem cell transplantation.

DETAILED DESCRIPTION:
This Phase 2 study will be conducted in patients with Hodgkin's disease, non-Hodgkin's lymphoma, multiple myeloma, or mantle cell lymphoma undergoing high-dose chemotherapy and autologous stem cell transplantation. Patients will be randomized to receive either LAD 11.25 mg 3 Month treatment or placebo and all patients will be vaccinated with KLH 6 months posttransplant. Patients will be evaluated to determine if the rate of immunologic recovery in the LAD group is enhanced compared with the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Must be female between the ages of 18 - 50 or if female > 50 years old have an estradiol concentration level >= 30 pg/mL and follicle stimulating hormone level < 40 mIU/mL, or male between the ages of 18-65 (inclusive).
2. Must have Hodgkin's disease, non-Hodgkin's lymphoma, multiple myeloma, or mantle cell lymphoma and be considered an appropriate candidate for hematopoietic stem cell transplant.

   1. Multiple myeloma patients should have had a partial or complete response to chemotherapy.
   2. Patients with Hodgkin's disease or non-Hodgkin's lymphoma who achieve a partial response to initial chemotherapy or first or second chemosensitive relapse, achieving a complete or partial response to salvage treatment. Patients in first remission with mantle cell lymphoma, or with intermediate or high grade lymphoma, presenting with high intermediate or high IPI (International Prognostic Index) scores are also eligible.
3. Must be seronegative for hepatitis C and HIV.
4. Must have received prior tetanus immunization
5. Must not have received prior KLH immunization.
6. Must have an ECOG performance status (PS) <= 1 or Karnofsky PS >= 70%.
7. Must have creatinine <= 2.0 mg/dL; ejection fraction > 45%; carbon monoxide diffusion in the lungs (DLCO) > 50% of predicted; serum bilirubin < 1.5 times the upper limit of normal unless Gilbert's syndrome, SGPT < 3 times normal value.
8. Must be more than 3 weeks from any prior surgery (except for central line placement) and have fully recovered from the effects of surgery.
9. Must have an absolute neutrophil count (ANC) >= 1,500 µL, platelet count >= 100,000/µL and hemoglobin >= 8.0 gm/dL within 21 days prior to randomization.
10. Must be able to return to the clinical site for follow-up visits.
11. Must be able to provide written consent.

Exclusion Criteria:

1. Must not have an uncontrolled life-threatening infection (or active infectious process requiring intravenous [IV] systemic medical therapy within 1 week prior to study enrollment).
2. Must not have a diagnosed or suspected schistosomiasis infection.
3. Must not have previously received hematopoietic stem cell transplantation.
4. Must not require a tandem transplant.
5. Must not be female with a positive pregnancy test, pregnant, or lactating and breast feeding, or wish to become pregnant during the course of the study. Must agree to use barrier method of contraception.
6. Must not be receiving estrogen or testosterone replacement therapy,phytoestrogen, phyto-testosterone, or oral contraceptives (patients may enroll if oral contraceptives are ceased prior to study entry), or have been administered Depo Provera within 3 months of entering the study.
7. Must not have had prior mediastinal or sternal radiation.
8. Must not have received any investigational drug other than antibiotics within 3 weeks prior to study drug administration or are scheduled to receive an investigational drug during the course of this study.
9. Must not have unstable cardiac arrhythmias, uncontrolled congestive heart failure, history of myocardial infarction (MI) or ischemia, stroke, or embolic events within 6 months before study start.
10. Must not have medical or psychiatric conditions that, in the opinion of the investigator, would compromise the patient's ability to participate in the study.
11. Must not be receiving or plan to receive palifermin (KGF).
12. Must not have a allergy to shellfish.
13. Must not have previously taken a GnRH analog within 18 months.
14. Must not be a woman who has undergone bilateral oophorectomy, or man with orchiectomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-02; Primary Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - St Louis, Missouri
  - New York, New York
  - Durham, North Carolina
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Leuprolide Acetate Depot (LAD) 11.25 mg 3 Month: Patients received 1 injection of LAD 11.25 mg every 3 months for a total treatment period of 9 months.
- Placebo: Patients received 1 injection of placebo every 3 months for a total treatment period of 9 months.
Period: Overall Study
Arm/Group | Leuprolide Acetate Depot (LAD) 11.25 mg 3 Month | Placebo
Started | 12 | 13
Completed | 6 (Patients who completed the entire 12 month study period) | 4 (Patients who completed the entire 12 month study period)
Not Completed | 6 | 9
Not completed — Adverse Event | 2 | 0
Not completed — Disease progression | 2 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Death | 1 | 0
Not completed — Started Chemotherapy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Leuprolide Acetate Depot (LAD) 11.25 mg 3 Month | Placebo | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49.0 (10.16) | 47.4 (7.04) | 48.2 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in IgM Response (Mcg/mL) Before Keyhole Limpet Hemocyanin (KLH) Vaccination at Month 6 and After KLH Vaccination at Month 7 in Patients Who Received LAD or Placebo
Description: Patients received a subcutaneous injection of KLH vaccine 1 month after subjects received the third injection of LAD or placebo. Serum immunoglobulin IgM antibodies were determined by enzyme-linked immunosorbent assay (ELISA). Baseline is defined as the IgM concentration before the KLH vaccination. Change from baseline was calculated as the IgM value postvaccination minus the IgM value at prevaccination.
Time Frame: Month 6 prevaccination (baseline) and Month 7 postvaccination
Population: Eight subjects from the LAD-treated arm and 5 subjects from the placebo-treated arm were assessed for IgM. These subjects received 3 doses of LAD or placebo, KLH vaccination, and had a blood collection suitable for analysis for primary endpoint although not all subjects completed the entire study.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Leuprolide Acetate Depot (LAD) 11.25 mg 3 Month | Placebo
Number analyzed (Participants) | 8 | 5
mcg/mL
  Mean IgM at baseline (mcg/mL) | 4.0 (3.8) [0.99 to 7.38] | 3.0 (2.8) [-0.16 to 1.84]
  Mean IgM change from baseline (mcg/mL) | 2.91 (2.07) | 0.57 (0.83)

2. Secondary Outcome: Mean Change From Baseline in T Cell Excision Circles (TREC) Per 100,000 CD4+ Cells to Final Visit in Patients Treated With LAD (11.25 mg) or Placebo After Transplant
Description: CD4+ cells are a type of T cell. T cells are produced in the thymus and thymic function can be determined by TREC. By counting the number of TRECs present (only 1 copy per cell) within a population of CD4 cells, an assessment of T cell recovery and immune response is obtained. Mayo Medical Clinic. http://www.mayomedicallaboratories.com/test-catalog/Clinical+and+Interpretive/87959. Accessed 17 MARCH 2010
  The change from baseline is defined as posttransplant TREC/100,000 CD4+ cells minus pretransplant TREC /100,000 CD4+ cells.
Time Frame: Pretransplant and posttransplant (Month 12)
Population: Nine subjects from the LAD-treated arm and 7 subjects from the placebo-treated arm were assessed for TREC per 100,000 CD4+ cells. These subjects received 3 doses of LAD or placebo, KLH vaccination, and had a blood collection suitable for analysis for primary endpoint although not all subjects completed the entire study.
Measure: Mean (Standard Deviation); unit: TREC /100,000 CD4+ cells
Arm/Group | Leuprolide Acetate Depot (LAD) 11.25 mg 3 Month | Placebo
Number analyzed (Participants) | 9 | 7
TREC /100,000 CD4+ cells
  Baseline TREC per 100,000 CD4+ cells | 67.524 (47.0863) | 173.712 (206.1733)
  Mean change in TREC from baseline to final visit | 522.321 (920.790) | -63.950 (235.561)
Statistical Analysis 1: Comparison: Leuprolide Acetate Depot (LAD) 11.25 mg 3 Month vs Placebo; The final on treatment values were included in the analysis; Test type: Superiority or Other; p = 0.125, ANOVA; The statistical method used for a 1-way ANOVA between treatment groups

3. Secondary Outcome: Mean Change From Baseline in TREC Per 100,000 CD8+ Cells to Final Visit in Patients Treated With LAD (11.25 mg) or Placebo After Transplant
Description: CD8+ cells are a type of T cell. T cells are produced in the thymus and thymic function can be determined by TREC. By counting the number of TRECs present (only 1 copy per cell) within a population of CD8+ cells, an assessment of T cell recovery and immune response is obtained. Mayo Medical Clinic. http://www.mayomedicallaboratories.com/test-catalog/Clinical+and+Interpretive/87959. Accessed 17 MARCH 2010
  The change from baseline is defined as posttransplant TREC/100,000 CD8+ cells minus pretransplant TREC /100,000 CD8+ cells.
Time Frame: Pretransplant and posttransplant (Month 12)
Population: Eight subjects from the LAD-treated arm and 5 subjects from the placebo-treated arm were assessed for TREC per 100,000 CD8+ cells. These subjects received 3 doses of LAD or placebo, KLH vaccination, and had a blood collection suitable for analysis for primary endpoint although not all subjects completed the entire study.
Measure: Mean (Standard Deviation); unit: TREC /100,000 CD8+ cells
Arm/Group | Leuprolide Acetate Depot (LAD) 11.25 mg 3 Month | Placebo
Number analyzed (Participants) | 9 | 7
TREC /100,000 CD8+ cells
  Baseline mean for TREC per 100,000 CD8+ cells | 181.673 (209.7599) | 364.414 (280.3465)
  Mean change in TREC from baseline to final visit | -10.811 (343.061) | -184.084 (282.405)
Statistical Analysis 1: Comparison: Leuprolide Acetate Depot (LAD) 11.25 mg 3 Month vs Placebo; The final on treatment values were included in the analysis; Test type: Superiority or Other; p = 0.299, ANOVA; The statistical method used for a 1-way ANOVA between treatment groups

4. Primary Outcome: Mean Change From Baseline in IgG1 Response (Mcg/mL) Before KLH Vaccination at Month 6 and After KLH Vaccination at Month 7 in Patients Who Received LAD or Placebo
Description: Patients received a subcutaneous injection of KLH vaccine 1 month after subjects received the third injection of LAD or placebo. Serum immunoglobulin IgG1 antibodies were determined by enzyme-linked immunosorbent assay (ELISA). Baseline is defined as the IgG1 concentration before the KLH vaccination. Change from baseline was calculated as the IgG1 value postvaccination minus the IgG1 value at baseline.
Time Frame: Month 6 prevaccination (baseline) and Month 7 postvaccination
Population: Eight subjects from the LAD-treated arm and 5 subjects from the placebo-treated arm were assessed for IgG1. These subjects received 3 doses of LAD or placebo, KLH vaccination, and had a blood collection suitable for analysis for primary endpoint although not all subjects completed the entire study.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Leuprolide Acetate Depot (LAD) 11.25 mg 3 Month | Placebo
Number analyzed (Participants) | 8 | 5
mcg/mL
  Mean IgG1 at baseline (mcg/mL) | 8.6 (9.1) | 10.8 (11.6)
  Mean IgG1 change from baseline (mcg/mL) | 46.16 (44.01) | 16.76 (28.15)

5. Primary Outcome: Mean Change From Baseline in Interferon Gamma Response (Spots/1 Million Cells) Before KLH Vaccination at Month 6 and After KLH Vaccination at Month 7 in Patients Who Received LAD or Placebo
Description: Patients received a subcutaneous injection of KLH vaccine 1 month after subjects received the third injection of LAD or placebo. Interferon gamma was determined by enzyme-linked immunosorbent spot-forming cell (ELISpot). Baseline is defined as the interferon gamma concentration obtained before the KLH vaccination. Change from baseline was calculated as the interferon gamma value postvaccination minus the interferon gamma value at baseline.
Time Frame: Month 6 prevaccination (baseline) and Month 7 postvaccination
Population: Six subjects from the LAD-treated arm and 5 subjects from the placebo-treated arm were assessed for interferon gamma. These subjects received 3 doses of LAD or placebo, KLH vaccination, and had a blood collection suitable for analysis for primary endpoint although not all subjects completed the entire study.
Measure: Mean (Standard Deviation); unit: spots/1 million cells
Arm/Group | Leuprolide Acetate Depot (LAD) 11.25 mg 3 Month | Placebo
Number analyzed (Participants) | 6 | 5
spots/1 million cells
  Mean interferon gamma at baseline | 0.2 (3.2) | -1.4 (3.2)
  Mean interferon gamma change from baseline | 2.09 (4.85) | 10.25 (11.41)

ADVERSE EVENTS:
Arm/Group | Leuprolide Acetate Depot (LAD) 11.25 mg 3 Month | Placebo
Serious Adverse Events (participants affected / at risk) | 6/12 | 4/13
Other Adverse Events (participants affected / at risk) | 7/12 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprolide Acetate Depot (LAD) 11.25 mg 3 Month (N=12) | Placebo (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Staphylococcal bacteremia (Infections and infestations) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprolide Acetate Depot (LAD) 11.25 mg 3 Month (N=12) | Placebo (N=13)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Hypogonadism (Endocrine disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Axillary pain (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Injection site swelling (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Edema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1
Central line infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Hemoglobin decreased (Investigations) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early because of slow enrollment. For the primary endpoint, changes from baseline within each treatment group were analyzed. Between treatment group comparisons were not performed because the sample size was too small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.